CLINICAL TRIAL: NCT04102267
Title: A Randomized, Phase 4 Study of the Efficacy, Safety, and Pharmacokinetics of Bupivacaine Administered as Liposomal Bupivacaine or Continuous Infusion Via Elastomeric Pump Following Unilateral Open Inguinal Herniorrhaphy
Brief Title: Extended Delivery of Bupivacaine Study in Herniorrhaphy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BUPI-501
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Analgesia
Keywords: herniorrhaphy; inguinal hernia; hernia; hernia surgery; postoperative pain
MeSH Terms: conditions — Agnosia; Hernia, Inguinal; Hernia; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal bupivacaine injection (Group 1) (Experimental): Liposomal bupivacaine 266 mg via injection
  Interventions: Drug: Bupivacaine liposome injectable suspension
- Bupivacaine HCl continuous infusion (Group 2) (Experimental): Bupivacaine HCl 300 mg via continuous infusion
  Interventions: Drug: Bupivacaine HCl without epinephrine via continuous infusion

INTERVENTIONS:
Drug: Bupivacaine liposome injectable suspension — Liposomal bupivacaine 266 mg via injection
  Arms: Liposomal bupivacaine injection (Group 1)
Drug: Bupivacaine HCl without epinephrine via continuous infusion — Bupivacaine HCl 300 mg via continuous infusion
  Arms: Bupivacaine HCl continuous infusion (Group 2)

SUMMARY:
This is a phase 4, randomized, open-label study of the efficacy, safety, and pharmacokinetics of bupivacaine administered as liposomal bupivacaine or continuous infusion via elastomeric pump following unilateral open inguinal herniorrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo a unilateral open inguinal herniorrhaphy with mesh under general anesthesia
* Has an American Society of Anesthesiologists Physical Status of I, II, or III
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile,or using acceptable contraceptives.

Exclusion Criteria:

* Had any prior inguinal hernia repair
* Has a planned concurrent surgical procedure
* Has other pre existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications
* Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.
* Has taken any NSAIDs within least 10 days prior to the scheduled surgery
* Has taken opioids within 24 hours prior to the scheduled surgery (3 days for long-acting)
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* Has initiated treatment with medications within 1 month prior to study drug administration that can impact pain control.
* Has been administered systemic steroids within 5 half-lives or 10 days prior to administration of study drug
* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments
* Has a known history of Hepatitis B, human immunodeficiency virus (HIV), or active Hepatitis C
* Has uncontrolled anxiety, psychiatric, or neurological disorder that, in the opinion of the Investigator, might interfere with study assessments
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse. Note: Subjects with a positive drug screen who are taking an allowed, prescribed medication that is known to result in a positive drug test (eg, amphetamine and dextroamphetamine for attention-deficit/hyperactivity disorder, benzodiazepine for anxiety disorder) may be eligible for participation in the study. Subjects taking medical marijuana are not allowed to participate in the study.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half-lives
* Has undergone 3 or more surgeries within 12 months
* Has a body mass index (BMI) >39 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Mean area under the curve (AUC) of the Numeric Rating Scale of pain intensity scores with activity (NRS-A) through 72 hours (AUC0-72) | 72 hours

SECONDARY OUTCOMES:
Total postoperative opioid consumption (in morphine equivalents) | 72 hours
Proportion of subjects who are opioid-free | 72 hours
Median time in hours to first opioid rescue medication | 72 hours
Mean AUC0-72 of the NRS-R pain intensity scores. | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States